CLINICAL TRIAL: NCT05365464
Title: hCG or Progesterone Effect on Unexplained Recurrent Pregnancy Loss
Brief Title: HOPE Trial hCG or Progesterone Effect on Recurrent Pregnancy Loss
Acronym: HOPE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator still working on protocol and not sure when it will be ready
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL3HOPE
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2021-08

CONDITIONS: Recurrent Pregnancy Loss Without Current Pregnancy
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Progesterone (Active Comparator): Women receive prometrium 200 mg qhs for up to 8 weeks
  Interventions: Drug: Progesterone Pill
- hCG (Active Comparator): A single shot of hCG (ovidril 250 ug) will be given as a subcutaneous injection 1 week after ovulation
  Interventions: Drug: hCG

INTERVENTIONS:
Drug: Progesterone Pill — Orally active progesterone
  Other Names: Prometrium
  Arms: Progesterone
Drug: hCG — Given by subcutaneous injection
  Other Names: Ovidril
  Arms: hCG

SUMMARY:
Up to half of all cases of recurrent pregnancy loss are unexplained (uRPL). Evidence points towards endometriosis and progesterone resistance as an underlying cause of uRPL. Previous non-RCT studies have suggested the luteal hCG provides a useful treatment for uRPL. We propose performing a randomized controlled trial to compare mid-luteal hCG with oral progesterone to prevent early pregnancy losses. the endpoint will be ongoing pregnancy and live birth rates. Equal numbers of patients will be randomized to each group.

DETAILED DESCRIPTION:
Fifty (50) patients with unexplained recurrent pregnancy loss, defined as 2 or more losses. Workup will exclude structural, genetic, hormonal, and anti-phospholipid syndrome-related causes of RPL. Women with unexplained RPL will be randomized to receive a mid-luteal injection of ovidril (250 ug) 1 week after ovulation vs prometrium (200 mg qhs) starting 4 days after ovulation. If pregnant, prometrium will be continued until 8 weeks of pregnancy. If pregnancy does not occur, subjects will be allowed to repeat this protocol for up to 3 cycles. Outcomes will be listed as "not pregnant", "biochemical pregnancy", "miscarriage" or "ongoing pregnancy" for each cycle. Endpoints of pregnant cycles will be compared for pregnancy rate, miscarriage rate, ongoing pregnancy rate and live birth rate.

ELIGIBILITY:
Inclusion Criteria:

* 2 first trimester losses
* unexplained recurrent pregnancy loss

Exclusion Criteria:

* Antiphospholipid syndrome
* uterine septum
* Asherman's syndrome
* Paternal or maternal genetic abnormalities (i.e. balanced translocation)
* Endocrine causes of RPL (thyroid, diabetes, hyperprolactinemia)

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnancy required
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Miscarriage | 4 to 11 weeks
  Loss of pregnancy before 11 weeks of pregnancy
Ongoing pregnancy | 8 weeks
  Successgful pregnancy beyond 8 weeks of gestation with a heart beat

SECONDARY OUTCOMES:
Live birth rate | 40 weeks
  Viable successful delivery of a life baby

IPD SHARING:
Plan to Share IPD: Undecided